CLINICAL TRIAL: NCT02808494
Title: Prospective Collection of Whole Blood Specimens of Subjects Diagnosed With Preeclampsia With Severe Features and/or Fetal Growth Restriction in Support of a Molecular Assay Development
Brief Title: Development of a Next Generation Sequencing (NGS) -Based Assay to Detect Preeclampsia Molecular Markers
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGH-014
Record Dates: First submitted 2016-04-26; First posted 2016-06-21 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Fetal Growth Restriction
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored for future assay development use.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Affected Group: Women with a diagnosis of preeclampsia with severe features and/or fetal growth restriction.
- Control/Unaffected Group: Women who do not have a diagnosis of preeclampsia with severe features and/or fetal growth restriction.

SUMMARY:
Sample Collection Study

DETAILED DESCRIPTION:
This is a limited prospective collection of whole blood samples from pregnant women with a diagnosis of preeclampsia with severe features and/or fetal growth restriction in addition to samples from a control group to aid in the development of a Next Generation Sequencing (NGS)-based assay to detect molecular markers associated with preterm preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older at enrollment
2. Pregnant women with a viable singleton gestation
3. Able to provide written, informed consent
4. Able to provide 20 mL of whole blood
5. Diagnosis of preeclampsia with severe features and/or diagnosis of fetal growth restriction.

   1. Preeclampsia with severe features is defined as:

      Proteinuria: Excretion of ≥300mg/24hr (24 hour collection) of protein or a timed excretion that is extrapolated to the 24 hour urine value or a protein/creatinine [both in mg/dL] ratio of at least 0.3 or a qualitative determination of (urine dipstick) of ≥1+ WITH Systolic BP ≥160mmHg or diastolic BP ≥110mmHg on at least 2 occasions 4 hours apart while on bedrest but before the onset of labor OR Systolic BP ≥160mmHg or diastolic BP ≥110mmHg on 1 occasion but before the onset of labor, if antihypertensive therapy is initiated due to severe hypertension OR New onset hypertension defined as: Systolic BP ≥140 mmHg or diastolic ≥90 mmHg with one or more of the following features: Thrombocytopenia (<100,000 plts/mL); impaired liver function (AST/ALT 2X ULN); newly developed renal insufficiency (serum creatinine >1.1mg/dL or a doubling of serum creatinine in the absence of other renal disease); pulmonary edema; new onset cerebral disturbances or scotomata
   2. Fetal Growth Restriction defined as:

   Estimated fetal weight by ultrasound at ≥ 19 0/7 weeks gestational age < 5%ile or 5-10%ile with abnormal umbilical artery Doppler examination (S/D ratio >95%ile for gestational age, absent end diastolic flow or reverse end diastolic flow)
6. Gestational age between 20 0/7 and 33 6/7 weeks determined by ultrasound and/or LMP per ACOG guidelines1. A subject diagnosed with preeclampsia without severe features prior to 33 6/7 weeks gestation and who is managed expectantly and develops severe features after 34 weeks may be included.

Exclusion Criteria:

1. Known malignancy
2. History of maternal organ or bone marrow transplant
3. Maternal blood transfusion in the last 8 weeks
4. Chronic hypertension diagnosed prior to current pregnancy
5. Type I, II or gestational diabetes
6. Fetal anomaly or known chromosome abnormality
7. Active labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Affected Group: Pregnant women diagnosed with preeclampsia with severe features or fetal growth restriction
  Control group: Pregnant women matched for gestational age to the Affected group above
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2016-03; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
cfRNA markers associated with preeclampsia with severe features and/or fetal growth restrictions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rhoa, MD, Study Director — Illumina, Inc.
Locations (10):
- United States (10):
  - Christiana Hospital, Newark, Delaware
  - Tufts Medical Center, Boston, Massachusetts
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers University, Piscataway, New Jersey
  - Virtua Materna-Fetal Medicine Specialists, Sewell, New Jersey
  - New York-Presbyterian/Queens, Flushing, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Winthrop University Hospital Clinical Trials Center, New York, New York
  - Drexel Medicine, Philadelphia, Pennsylvania
  - The University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Munchel S, Rohrback S, Randise-Hinchliff C, Kinnings S, Deshmukh S, Alla N, Tan C, Kia A, Greene G, Leety L, Rhoa M, Yeats S, Saul M, Chou J, Bianco K, O'Shea K, Bujold E, Norwitz E, Wapner R, Saade G, Kaper F. Circulating transcripts in maternal blood reflect a molecular signature of early-onset preeclampsia. Sci Transl Med. 2020 Jul 1;12(550):eaaz0131. doi: 10.1126/scitranslmed.aaz0131. PMID 32611681